CLINICAL TRIAL: NCT00042822
Title: A Pilot Study Of FR901228, Or Depsipeptide (NSC #630176) For Adult Patients With Advanced Hematologic Cancers
Brief Title: FR901228 in Treating Patients With Myelodysplastic Syndrome, Acute Myeloid Leukemia, or Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000069473; MSKCC-00116; NCI-1715
Record Dates: First submitted 2002-08-05; First posted 2003-01-27 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2009-12

CONDITIONS: Leukemia; Lymphoma; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms
Keywords: recurrent adult acute myeloid leukemia; refractory anemia with excess blasts; refractory anemia with excess blasts in transformation; chronic myelomonocytic leukemia; recurrent grade 3 follicular lymphoma; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; untreated adult acute myeloid leukemia; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; atypical chronic myeloid leukemia, BCR-ABL1 negative; myelodysplastic/myeloproliferative neoplasm, unclassifiable; adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with t(15;17)(q22;q12)
MeSH Terms: conditions — Leukemia; Lymphoma; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Leukemia, Myeloid, Acute; Anemia, Refractory, with Excess of Blasts; Leukemia, Myelomonocytic, Chronic; Lymphoma, Follicular; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Myeloproliferative Disorders; Congenital Abnormalities | interventions — romidepsin

INTERVENTIONS:
Drug: romidepsin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of FR901228 in treating patients who have myelodysplastic syndrome, acute myeloid leukemia, or non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the pattern of adverse clinical experience in patients with myelodysplastic syndrome, acute myeloid leukemia, or intermediate-grade or follicular non-Hodgkin's lymphoma treated with FR901228 (depsipeptide).
* Determine the disease response in patients treated with this drug.
* Determine the pharmacokinetic and pharmacodynamic correlates of this drug, including measurement of serum plasma levels, H3 and H4 acetylation, apoptosis induction, differentiation, and multidrug-resistant (MDR) phenotype expression in these patients.

OUTLINE: Patients receive FR901228 (depsipeptide) IV over 4 hours on days 1 and 5. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients are followed monthly.

PROJECTED ACCRUAL: A total of 12 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* One of the following diagnoses:

  * Histologically confirmed refractory or relapsed acute myeloid leukemia (AML)

    * Failed anthracycline-based chemotherapy
    * Ineligible for or refused allogeneic stem cell transplantation
  * Elderly patients with newly diagnosed AML

    * Ineligible for or refused standard chemotherapy
  * Histologically confirmed high-risk myelodysplastic syndromes

    * Eligible subtypes include:

      * Refractory anemia with excess blasts (RAEB)
      * RAEB in transformation
      * Chronic myelomonocytic leukemia
    * Ineligible for or refused allogeneic bone marrow transplantation
  * Histologically confirmed intermediate-grade non-Hodgkin's lymphoma (NHL)

    * Relapsed after high-dose therapy OR
    * Ineligible for allogeneic or autologous stem cell transplantation
    * Evaluable lesions by radiologic study or physical examination
  * Histologically confirmed follicular NHL

    * Progressed after anthracycline-based chemotherapy and rituximab
    * Evaluable lesions by radiologic study or physical examination NOTE: A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 60-100%

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Bilirubin no greater than 1.5 mg/dL (unless due to Gilbert's syndrome)
* SGOT and SGPT less than 2 times upper limit of normal

Renal

* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance at least 60 mL/min

Cardiovascular

* Cardiac ejection fraction greater than 50%
* No cardiac hypertrophy
* No known conduction heart disease
* No New York Heart Association class III or IV heart disease that would make it difficult to assess patient during study participation
* No significant prior heart disease
* No significant prior secondary or tertiary heart block
* No significant prior atrial or ventricular arrhythmia requiring therapeutic intervention or antiarrhythmics for rate control

Pulmonary

* No severe debilitating pulmonary disease that would make it difficult to assess patient during study participation

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 1 month after study participation
* Potassium ≥ 4.0 mmol/L (supplementation allowed)
* Magnesium ≥ 2.0 mg/dL (supplementation allowed)
* No other concurrent active malignancy except basal cell skin cancer
* No other concurrent significant co-morbidity that would make it difficult to assess patient during study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* At least 2 weeks since prior epoetin alfa or filgrastim (G-CSF)
* At least 4 weeks since prior cytokines
* No concurrent immunotherapy

Chemotherapy

* See Disease Characteristics
* At least 4 weeks since prior systemic chemotherapy
* No other concurrent chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* At least 4 weeks since prior radiotherapy
* No concurrent radiotherapy

Surgery

* Not specified

Other

* No other concurrent investigational agents
* No concurrent drugs that may prolong the QTc interval

  * FR901228 (depsipeptide) may be administered after a 5-half-life washout period following the use of these drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-05; Primary Completion 2005-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Klimek, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Result] Klimek VM, Fircanis S, Maslak P, Guernah I, Baum M, Wu N, Panageas K, Wright JJ, Pandolfi PP, Nimer SD. Tolerability, pharmacodynamics, and pharmacokinetics studies of depsipeptide (romidepsin) in patients with acute myelogenous leukemia or advanced myelodysplastic syndromes. Clin Cancer Res. 2008 Feb 1;14(3):826-32. doi: 10.1158/1078-0432.CCR-07-0318. PMID 18245545